CLINICAL TRIAL: NCT01746524
Title: Prospective, Single Arm Multiconfiguration Investigation to Assess Functional Performance of Attune™ Primary Total Knee Arthroplasty System
Brief Title: Prospective, Multiconfiguration Study to Assess Functional Performance of Primary Total Knee Arthroplasty System
Acronym: 10004
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 10004
Record Dates: First submitted 2012-12-05; First posted 2012-12-11 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; Replacement; Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CR FB: Subjects receiving Cruciate Retaining Fixed Bearing configuration of ATTUNE Primary Knee Implant
  Interventions: Device: ATTUNE Primary Total Knee Arthroplasty
- PS FB: Subjects receiving Posterior Stabilized Fixed Bearing configuration of ATTUNE Primary Knee Implant
  Interventions: Device: ATTUNE Primary Total Knee Arthroplasty
- CR RP: Subjects receiving Cruciate Retaining Rotating Platform configuration of ATTUNE Primary Knee Implant
  Interventions: Device: ATTUNE Primary Total Knee Arthroplasty
- PS RP: Subjects receiving Posterior Stabilized Rotating Platform configuration of ATTUNE Primary Knee Implant
  Interventions: Device: ATTUNE Primary Total Knee Arthroplasty

INTERVENTIONS:
Device: ATTUNE Primary Total Knee Arthroplasty — Patients will undergo a primary, cemented total knee replacement using one of the four configurations of the Attune knee (CR FB, PS FB, CR RP, PS RP).

SUMMARY:
This post-marketing investigation will evaluate the functional knee performance of Subjects who have undergone primary total knee arthroplasty (TKA). Data from Subjects who receive one of four contemporary knee configurations will be pooled to establish a contemporary dataset.

The primary objective of this study is to evaluate the pre-operative (approximately -90 to -1 day before surgery) to minimum one year (approximately 304 to 668 days) postoperative functional performance improvement for the Attune™ primary, cemented TKA system as measured by the activities of daily living (ADL)subscore of the Knee Osteoarthritis Outcomes Score (KOOS)questionnaire (KOOS-ADL sub-score). This will be carried out for all four implant configurations: cruciate retaining fixed bearing (Attune™ CR FB), cruciate retaining rotating platform (Attune™ CR RP), posterior stabilized fixed bearing (Attune™ PS FB), and posterior stabilized rotating platform (Attune™ PS RP).

DETAILED DESCRIPTION:
The study is designed as a prospective, single arm stratified, multi-center investigation.

Approximately 20 study sites, worldwide, will enroll 1040 subjects (1040 knees). Each study is expected to enroll approximately 52 subjects (approximately 52 knees). An additional 10 subjects per site may be recruited at sites which have Sub-Investigators participating in the study. Cohort reallocation is permitted. There will be no control group. One thousand and forty (1040)Subjects will be stratified into 4 subgroups of 260: cruciate retaining fixed bearing(CR FB), posterior stabilized fixed bearing (PS FB), cruciate retaining rotating platform (CR RP), and posterior stabilized rotating platform (PS RP). Treatment assignment in this study is not randomized.

Each site will only enroll patients in one of the four knee configuration sub-groups most commonly used as their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 22 and 80 years, inclusive.
* Subject was diagnosed with NIDJD.
* Subject is a suitable candidate for cemented primary TKA using the devices described in the Clinical Investigation Plan (CIP)with either resurfaced or non-resurfaced patellae.
* Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to DePuy.
* Subject is currently not bedridden.
* Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and co-operate with investigational procedures.
* Subject must be comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the PROs in the CIP.
* The devices specified in this CIP were implanted.

Exclusion Criteria:

* The Subject is a woman who is pregnant or lactating.
* Contralateral knee has already been enrolled in this study.
* Subject had a contralateral amputation.
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently experiencing radicular pain from the spine.
* Subject has participated in an IDE/IND clinical investigation with an investigational product in the last three months.
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject is a known drug or alcohol abuser or has a psychological disorder that could affect their ability to complete patient reported questionnaires.
* Subject was diagnosed with fibromyalgia that is currently being treated with prescription medication.
* Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).
* Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the PROs in the CIP.
* Subject has a medical condition with less than 2 years of life expectancy.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female Subjects, age 22-80 years, inclusive, with Non-inflammatory Degenerative Joint Disease (NIDJD) who are suitable candidates for primary TKA using the Attune system.
Sampling Method: Non-Probability Sample
Enrollment: 1138 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) activities of daily living (ADL) sub-score change from baseline. | One year or later (approximately 304 days or later)
  The KOOS ADL will be measured before surgery and at a minimum 1 year after surgery. The KOOS is a patient self-administered questionnaire that consists of 42 questions. The KOOS consists of 5 subscales; pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee-related quality of life. Each question has 5 Likert-like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The change from baseline is the minimum 1 year (approximately 304 to 668 days) measurement minus the baseline measurement.

SECONDARY OUTCOMES:
Patient Reported Outcome: Oxford Knee Score (OKS) | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  The Oxford Knee Score (OKS) is a patient self-administered 12-item questionnaire with each question having 5 Likert- like response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OKS measures pain and general activities of daily living.
Patient Reported Outcome: Pre-surgical/Post-surgical Patient's Knee Implant Performance (PKIP) | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  The Pre Surgical and/or Post-surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient self-administered questionnaire that consists of 25 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likert- like response option.
Patient Report Outcome: EuroQol 5D 3L questionnaire (EQ-5D-3L) | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  EuroQol 5D 3L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Type and Frequency of Adverse Events (AEs) for all enrolled subjects | < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  All Serious AEs must be reported to Sponsor. All device-related or procedure-related adverse events must be reported to Sponsor.
Evaluate primary cemented fixation through zonal radiographic analysis post-operatively | minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  Radiographs will be reviewed by an independent radiographic reviewer (IRR). Data from the IRR radiographic evaluations will be used for determination of radiographic success criteria.
Incidence of post-operative anterior knee pain and symptomatic/asymptomatic crepitus | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  The Anterior Knee Pain and Crepitus questionnaire will be used. It is a 2 part questionnaire that is patient-self administered. The crepitus questions include frequency of crepitus and whether or not crepitus is symptomatic. The anterior knee pain contains 2 questions that collect frequency of pain and location of pain.
Evaluate surgeon learning curve on clinical and functional outcomes | < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  Each surgeon will implant devices into the first 10 Subjects which will be considered as 'learning curve cases'; these learning curve cases will not be pooled with post-learning curve cases unless learning curve analyses indicate that there is not a significant learning curve with regard to clinical or functional Subject outcomes.
Evaluate the impact of ligament balancing surgical technique on functional performance | Operatively (Day 0 - Date of Surgery)
  Description of the Subject's surgical procedure including such items as surgical approach and ligament balancing will be evaluated.
Psychometric Properties of the Patient Knee Implant Performance (PKIP)questionnaire | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  The Pre and Post-Surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient self-administered questionnaire that consists of 25 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likert- like response option.
Evaluate the functional outcome of patella resurfacing and non-resurfacing | < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  An exploratory comparison of results between knees with patella resurfacing versus knees without resurfacing will be conducted. A comparison of KOOS, PKIP, OKS, Knee Society (AKS), anterior knee pain incidence, and crepitus will be conducted.
Evaluate changes in femoral component and tibial component alignment | < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  Radiographs will be reviewed by an independent radiographic reviewer (IRR) in order to minimize bias of radiographic outcomes. Data from the IRR radiographic evaluations will be used to evaluate femoral and tibial component alignment over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S, Ismail, MS, CCRP, Study Director — DePuy Orthopaedics
Locations (20):
- United States (9):
  - Orthopaedic Specialty Institute, Orange, California
  - UCSD Medical Center, San Diego, California
  - Orhopaedic Center of the Rockies, Fort Collins, Colorado
  - The Arthroplasty Foundation, Louisville, Kentucky
  - Hip and Knee Research of Nevada, Las Vegas, Nevada
  - Dartmouth Medical School/Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cardinal Orthopaedic Institute, Columbus, Ohio
  - Anderson Orthopaedic Research Institute, Alexandria, Virginia
  - Swedish Orthopedic Institute, Seattle, Washington
- Australia (4):
  - Sutherland Hospital, Caringbah, New South Wales
  - Hornsby Ku-ring-gai Hospital, Hornsby, New South Wales
  - Wakefield Orthopaedic Clinic, Adelaide, South Australia
  - Freemantle Hospital, Crawley, Western Australia
- Ascot Hospital, Auckland, New Zealand
- United Kingdom (6):
  - Queen Margaret Hospital, Dunfermline, Fife
  - The Royal Surrey County Hospital, Guildford, Surrey
  - Princess Alexandra Hospital, Harlow
  - University Hospital Llandough, Llandough
  - James Cook University Hospital, Middlesbrough
  - Clifton Park NHS Treatment Centre, York

REFERENCES:
- [Derived] Hamilton WG, Brenkel IJ, Barnett SL, Allen PW, Dwyer KA, Lesko JP, Kantor SR, Clatworthy MG. Comparison of Existing and New Total Knee Arthroplasty Implant Systems From the Same Manufacturer: A Prospective, Multicenter Study. J Am Acad Orthop Surg Glob Res Rev. 2021 Dec 15;5(12):e21.00136. doi: 10.5435/JAAOSGlobal-D-21-00136. PMID 34908561